CLINICAL TRIAL: NCT03216811
Title: Nutraceutical Compound to Optimize Cholesterol, Endothelial and Inflammatory Parameters in Subjects With Hypercholesterolemia and Low to Moderate Cardiovascular Risk: the NIRVANA Study
Brief Title: Nutraceutical in Cardiovascular Primary Prevention
Acronym: NIRVANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, Interventional Cardiologist, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170598
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Subjects that meet the inclusion/exclusion criteria and have provided informed consent will undergo a 4-week period of lifestyle advice and changes. If, after the 4 weeks, LDL values are confirmed above the established cutoffs, the subjects receive CARDIOVIS COLESTEROLO 3 mg for 8 weeks. After the 8-week treatment period, all biological paprameters will be reassessed. Finally, a last blood samples to assess a potential rebound effect after nutraceutical suspension is collected 4 weeks after the treatment stop.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutraceutical (Experimental): after 4 weeks of lifestyle advice and changes, all subjects will receive for 8 weeks the administration of CARDIOVIS COLESTEROLO 3 mg, a nutraceutical compound containing containing red rice fermented with Monascus purpureus titrated with 3% monacolin K, hydrol mixture of olive fruit titrated with vitamin E, Coenzyme Q10 and polymethoxyflavones
  Interventions: Drug: nutraceutical

INTERVENTIONS:
Drug: nutraceutical — 8-week administration of nutraceutical compound

SUMMARY:
Nutraceuticals have attracted interest as possible approach to be associated with lifestyle changes for lowering plasma cholesterol levels in patients with moderate hypercholesterolemia. Ruscica and colleagues showed that a 8-weeks treatment with a nutraceutical combination containing red yeast rice extract, berberine, policosanol, astaxanthin, coenzyme Q10, and folic acid was able to reduce significantly total cholesterol (-12.8%) and low-density lipoprotein-cholesterol (-21.1%) [11]. These nutraceutical compounds exert their lipid-lowering effect through different ways, like the inhibition of the hydroxymethylglutaryl coenzyme A (CoA) enzyme, increasing the hepatic expression of low density lipoprotein (LDL) receptor and the LDL degradation via enhanced hepatic binding and internalization. In addition, they up regulate the numbers and function of circulating endothelial progenitor cells increasing nitric oxide (NO) production. The purpose of the present study was to assess the effectiveness of CARDIOVIS COLESTEROLO 3 mg (containing red rice fermented with Monascus purpureus titrated with 3% monacolin K, hydrol mixture of olive fruit titrated with vitamin E, Coenzyme Q10 and polymethoxyflavones) in terms of cholesterol, endothelial and inflammatory parameters reduction.

DETAILED DESCRIPTION:
Epidemiology. Cardiovascular disease (CVD) is the most common cause of death globally: an estimated 17.5 million people died from CVD in 2012, representing 31% of all global deaths. Of these deaths, an estimated 7.4 million were due to coronary heart disease and 6.7 million were due to stroke. Consistent evidences suggest that a large proportion of CVD incidence could be prevented by lifestyle modifications.

Atherosclerosis, hypercholesterolemia, inflammation and endothelial dysfunction Atherosclerosis covers a central rule in cardiovascular diseases. This process can be promoting by several risk factors, all related with endothelial dysfunction, as hypercholesterolemia, diabetes, cigarette smoking and arterial hypertension that acting as negative stimuli lead to a prothrombotic pathway by proinflammatory-induced cytokines and chemokine's production. Furthermore endothelial cells exposed to hypercholesterolemia are inhibited by the downregulation of extracellular nitric oxide synthase (eNOS) in the release of endothelium-derived relaxing factor, thus the benefits of lowering cholesterol are not only related to its primary implication in the atherosclerosis process, but also by the improvement of the endothelial function.

Cardiovascular risk (systematic coronary risk evaluation, SCORE). Current guidelines recommend the cardiovascular risk estimation, using a risk estimation system such as SCORE, for adults >40 years of age, unless they are automatically categorized as being at high-risk or very high-risk based on documented cardiovascular disease, diabetes mellitus, or kidney disease. A patient is defined at low to moderate risk when the cardiovascular risk is below 5%. Interventional strategies for hypercholesterolemia. The current guidelines recommendations for the management of hypercholesterolemia according cardiovascular risk are reported below in the Table. In addition to lifestyle advice, drugs may be considered in patients at low risk if LDL values are ≥ 190 mg/dl and in patients at moderate risk if LDL values are ≥ 100 mg/dl.

Nutraceuticals Several studies have assessed the effect of dietary interventions on risk factors for CVDs, but there is often lack effectiveness in the long term, mainly due to poor compliance. Research has thus turned its attention to nutraceuticals, nutrients that have the ability to modulate physiological and pathophysiological molecular mechanisms, resulting in favorable health outcomes. Nutraceuticals enhance cardiovascular health through several metabolic pathways as via promoting vasodilatory, anti-atherogenic, antioxidant, antithrombotic and anti-inflammatory effects]. Of note the extracts of red yeast rice explicate a lowering lipid action through monacolins, a family of naturally occurring statins, especially monacolin K, that is an inhibitor of the hydroxymethylglutaryl-CoA enzyme. Several trials of its possible lipid-lowering effects have been conducted and a meta-analysis [10] assesses the effectiveness and safety of preparations on lipid modification. Nutraceuticals have attracted interest as possible approach to be associated with lifestyle changes for lowering plasma cholesterol levels in patients with moderate hypercholesterolemia. Ruscica and colleagues showed that a 8-weeks treatment with a nutraceutical combination containing red yeast rice extract, berberine, policosanol, astaxanthin, coenzyme Q10, and folic acid was able to reduce significantly total cholesterol (-12.8%) and low-density lipoprotein-cholesterol (-21.1%). These nutraceutical compounds exert their lipid-lowering effect through different ways, like the inhibition of the hydroxymethylglutaryl-CoA enzyme, increasing the hepatic expression of LDL receptor and the LDL degradation via enhanced hepatic binding and internalization. In addition, they up regulate the numbers and function of circulating endothelial progenitor cells increasing NO production. The purpose of the present study was to assess the effectiveness of CARDIOVIS COLESTEROLO 3 mg (containing red rice fermented with Monascus purpureus titrated with 3% monacolin K, hydrol mixture of olive fruit titrated with vitamin E, Coenzyme Q10 and polymethoxyflavones) in terms of cholesterol, endothelial and inflammatory parameters reduction.

This is a prospective, single-center, and phase IIb study evaluating the effectiveness of CARDIOVIS COLESTEROLO 3 MG in improving cholesterol, endothelial and inflammatory parameters. Subjects that meet the inclusion criteria and have provided informed consent will be assigned to receive a daily oral dose of CARDIOVIS COLESTEROLO 3 mg. Before the treatment with CARDIOVIS COLESTEROLO 3 mg all subjects undergo a 4-week period of lifestyle advice and changes. If, after the 4 weeks, LDL values are confirmed above the established cutoffs, the subjects receive CARDIOVIS COLESTEROLO 3 mg. Finally, a last blood samples to assess a potential rebound effect after nutraceutical suspension is collected 4 weeks after the treatment stop.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years; Ability to provide informed written consent and to participate in the 16 weeks follow-up period And one of the following criteria

* Cardiovascular risk (SCORE) <1% and LDL levels ≥ 190 mg/dl (confirmed after a 4-week period of life style changes)
* Cardiovascular risk (SCORE) 1% to <5% and LDL levels ≥ 100 mg/dl (confirmed after a 4- week period of life style changes)

Exclusion Criteria:

Chronic liver disease Renal disease (creatinine clearance <60 mg/dl) Intolerance to nutraceutical compounds Thyroid disease Alcohol consumption >40 g/die Treatment with lipid lowering products in the previous 4 weeks Known coronary artery disease (CAD) or cerebrovascular disease Cardiovascular risk (SCORE) ≥5%

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
LDL | 8 weeks
  blood values of low density lipoprotein

SECONDARY OUTCOMES:
triglycerides | 8 weeks
  blood values of triglycerides
total cholesterol | 8 weeks
  blood values of total cholesterol
oxidized LDL | 8 weeks
  blood values of oxidized LDL
HDL | 8 weeks
  blood values of high density lipoprotein
rate of apoptosis | 8 weeks
  rate of apoptosis in human umbilical vein endothelial cells treated with subject's serum
radical oxygen species (ROS) | 8 weeks
  blood values of ROS generation
nitric oxide (NO) | 8 weeks
  NO generation in human umbilical vein endothelial cells treated with subject's serum

OTHER OUTCOMES:
creatine phosphate kinase (CPK) | 8 weeks
  blood values of CPK

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cimaglia, Dr, Principal Investigator — University Hospital of Ferrara; Francesco Vitali, Dr, Principal Investigator — University Hospital of Ferrara
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cimaglia P, Vieceli Dalla Sega F, Vitali F, Lodolini V, Bernucci D, Passarini G, Fortini F, Marracino L, Aquila G, Rizzo P, Ferrari R, Campo G. Effectiveness of a Novel Nutraceutical Compound Containing Red Yeast Rice, Polymethoxyflavones and Antioxidants in the Modulation of Cholesterol Levels in Subjects With Hypercholesterolemia and Low-Moderate Cardiovascular Risk: The NIRVANA Study. Front Physiol. 2019 Mar 11;10:217. doi: 10.3389/fphys.2019.00217. eCollection 2019. PMID 30914970